CLINICAL TRIAL: NCT02704325
Title: Phase I Gene Transfer Clinical Trial for Duchenne Muscular Dystrophy Using rAAVrh74.MCK.GALGT2
Brief Title: Gene Transfer Clinical Trial for Duchenne Muscular Dystrophy Using rAAVrh74.MCK.GALGT2
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kevin Flanigan (Other)
Responsible Party: Sponsor-Investigator, Kevin Flanigan, Professor of Pediatrics, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALGT2 for DMD
Record Dates: First submitted 2015-12-23; First posted 2016-03-10 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a dose escalation trial that will begin with the minimal efficacious dose as determined by preclinical studies and approved by the FDA. During the course of the trial, if safety is shown the dose will be escalated according to the clinical protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GALGT2 Viral Vector (Experimental): Dose: 1E12 vg (total dose) (n=3) of rAAVrh74.MCK.GALGT2 vs Placebo (Saline). All participants will receive rAAVrh74.MCK.GALGT2 in the right or the left EDB muscle and receive Saline in the opposite EDB muscles. The investigator will not know which side will receive rAAVrh74.MCK.GALGT2 vs Saline until after the trial is over. At the end of the trial the investigator will be unblinded.
  Interventions: Biological: rAAVrh74.MCK.GALGT2
- Saline (Experimental): Dose: 1E12 vg (total dose) (n=3) of rAAVrh74.MCK.GALGT2 vs Placebo (Saline). All participants will receive rAAVrh74.MCK.GALGT2 in the right or the left EDB muscle and receive Saline in the opposite EDB muscles. The investigator will not know which side will receive rAAVrh74.MCK.GALGT2 vs Saline until after the trial is over. At the end of the trial the investigator will be unblinded.
  Interventions: Other: PLACEBO (Saline)

INTERVENTIONS:
Biological: rAAVrh74.MCK.GALGT2 — Direct intramuscular injection of rAAVrh74.MCK.GALGT2 transferred to the extensor digitorum brevis muscle (EDB) of one foot and the other side receiving saline alone.
  Arms: GALGT2 Viral Vector
Other: PLACEBO (Saline) — Direct intramuscular injection of rAAVrh74.MCK.GALGT2 transferred to the extensor digitorum brevis muscle (EDB) of one foot and the OTHER side receiving saline alone.
  Arms: Saline

SUMMARY:
The proposed clinical trial study of rAAVrh74.MCK.GALGT2 for duchenne muscular dystrophy (DMD) patients that will involve direct intramuscular injection to the extensor digitorum brevis muscle (EDB).

DETAILED DESCRIPTION:
This is a phase I safety and tolerability study. Three DMD subjects will receive bilateral injections into the EDB muscle, with one EDB receiving the GALGT2 vector (rAAVrh74.MCK.GALGT2) and the other side receiving saline alone (assigned in a randomized fashion). Three subjects will receive a single gene transfer dose of 1E12 vector genomes, and patients and investigators will be blinded as to which muscle is injected with vector. Muscle biopsies will be performed at three months (12 weeks) in two subjects and at 1.5 months (6 weeks) in one subject and evaluated blindly for the expression of the GALGT2 transgene.

ELIGIBILITY:
Inclusion Criteria:

* Nonambulant subjects, age 9 or older
* Confirmed mutation in the DMD gene using a clinically accepted technique that completely defines the mutation
* A magnetic resonance image of the EDB showing preservation of sufficient muscle mass to permit transfection
* Males of any ethnic group will be eligible
* Ability to cooperate with all study procedures
* Willingness of sexually active subjects with reproductive capacity to practice reliable method of contraception (If appropriate).
* Stable dose of corticosteroid therapy (including either prednisone or deflazacort and their generic forms) for 12 weeks prior to gene transfer

Exclusion Criteria:

* Active viral infection based on clinical observations.
* The presence of a DMD mutation without weakness or loss of function
* Symptoms or signs of cardiomyopathy, including:
* Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
* Echocardiogram with ejection fraction below 40%
* Serological evidence of HIV infection, or Hepatitis A, B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥ 20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Subjects with rAAVrh74 binding antibody titers ≥ 1:400 as determined by ELISA immunoassay
* Presence of circulating anti-Sda antibodies as determined by study approved laboratory.
* Abnormal laboratory values in the clinically significant range, based upon normal values in the Nationwide Children's Hospital Laboratory

Min Age: 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Treatment related toxicities | 2 years
  Based on the development of unacceptable toxicity defined as the occurrence of any one Grade III or higher treatment-related toxicities.

SECONDARY OUTCOMES:
Expression of GALGT2 demonstrated with anti-CT epitope antibodies. | 6 or 12 weeks
GALGT2 protein expression quantified by western blot and assessed by densitometry | 6 or 12 weeks
Transduction efficiency measured by qPCR of the GALGT transgene from muscle, and expressed as vector genomes normalized to a genomic single-copy control. | 6 or 12 weeks
Number of fibers containing central nuclei compared between muscles by paired t-tests | 6 or 12 weeks
Dystrophin expression demonstrated with antibodies to N-terminal, C-terminal, and rod domains | 6 or 12 weeks
Utrophin expression | 6 or 12 weeks
Leukocyte markers including CD45, CD3, CD4, CD8, and MAC 387 | 6 or 12 weeks
Muscle will be examined for histological appearance | 6 or 12 weeks
Antibodies to rAAVrh74 along with PBMC ELISpots to both rAAVrh74 capsid and GALGT protein will be evaluated at different time points during the study | 6 or 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Flanigan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Chicoine LG, Rodino-Klapac LR, Shao G, Xu R, Bremer WG, Camboni M, Golden B, Montgomery CL, Shontz K, Heller KN, Griffin DA, Lewis S, Coley BD, Walker CM, Clark KR, Sahenk Z, Mendell JR, Martin PT. Vascular delivery of rAAVrh74.MCK.GALGT2 to the gastrocnemius muscle of the rhesus macaque stimulates the expression of dystrophin and laminin alpha2 surrogates. Mol Ther. 2014 Apr;22(4):713-24. doi: 10.1038/mt.2013.246. Epub 2013 Oct 22. PMID 24145553
- [Background] Martin PT, Xu R, Rodino-Klapac LR, Oglesbay E, Camboni M, Montgomery CL, Shontz K, Chicoine LG, Clark KR, Sahenk Z, Mendell JR, Janssen PM. Overexpression of Galgt2 in skeletal muscle prevents injury resulting from eccentric contractions in both mdx and wild-type mice. Am J Physiol Cell Physiol. 2009 Mar;296(3):C476-88. doi: 10.1152/ajpcell.00456.2008. Epub 2008 Dec 24. PMID 19109526